CLINICAL TRIAL: NCT06111391
Title: Patient Satisfaction , Prosthetic Complication and Clinical Outcomes of PEEK Composite Versus Titanium Zirconium Maxillary Fixed Full Arch Prosthetic Opposing Mandibular Distal Extension Partial Denture
Brief Title: Patient Satisfaction , Prosthetic Complications and Clinical Outcomes of PEEK Composite Versus Titanium Zirconium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A27080622
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-02

CONDITIONS: Patient Satisfaction; Prosthetic Complication; Clinical Outcomes
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maxillary titanium zirconium full arch fixed prosthesis (Active Comparator): maxillary titanium zirconium full arch fixed prosthesis and mandibular distal extension partial denture.
  Interventions: Device: Osstell® device (Integration Diagnostics Ltd.).
- maxillary peek composite full arch fixed prosthesis (Active Comparator): maxillary peek composite full arch fixed prosthesis and mandibular distal extension partial denture.
  Interventions: Device: Osstell® device (Integration Diagnostics Ltd.).

INTERVENTIONS:
Device: Osstell® device (Integration Diagnostics Ltd.). — After trans-mucosal abutments were removed and the smart pegs were attached to the fixtures, resonance frequency analysis was done to assess implant stability.The implant stability quotient (ISQ) was used to quantify stability via the Osstell® device (Integration Diagnostics Ltd.).

SUMMARY:
This study aimed to evaluate patient satisfaction (VAS) , prosthetic outcomes and clinical outcomes of polyether ether ketone (PEEK) Versus Titanium Zirconium fixed prostheses supported by six maxillary implants and opposed by distal extension removable partial denture.

DETAILED DESCRIPTION:
thirty patients were selected for this study from a previous study who have already received previous implants in the maxillary arch. The patients were divided into two groups: Group1 received maxillary titanium zirconium full arch fixed prosthesis and mandibular distal extension partial denture, Group 2 received maxillary PEEK composite full arch fixed prosthesis and mandibular distal extension partial denture Patient satisfaction was evaluated using visual analogue scale (VAS) after one year months , Prosthetic complications were measured on the patient and implant levels after one year

ELIGIBILITY:
Inclusion Criteria:

Normal jaw relation Good oral hygiene Patient with class I or class II inter-rach space in order to have sufficient restoration space to construct FP3 prosthesis.

Exclusion Criteria:

Patients with TMJ disorder and heavy smokers for more than 10 cigarettes per day.

Uncooperative patient. Unfavorable occlusion. Limited restoration space (less than 12 mm).

Ages: 58 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
implant stability | 12 months
  After transmucosal abutments were removed and the smart pegs were attached to the fixtures, resonance frequency analysis was done to assess implant stability.The implant stability quotient (ISQ) was used to quantify stability via the Osstell® device (Integration Diagnostics Ltd.).

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Aboelez, Phd, Study Director — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Wu P, Liu HL, Zhang L, Liu LP, Ma CF, Chen JH. Polyetheretherketone versus titanium CAD-CAM framework for implant-supported fixed complete dentures: a retrospective study with up to 5-year follow-up. J Prosthodont Res. 2022 Apr 27;66(2):279-287. doi: 10.2186/jpr.JPR_D_20_00142. Epub 2021 Sep 30. PMID 34588401